CLINICAL TRIAL: NCT04248088
Title: Getting Into Light Exercise for Patients With Heart Failure
Acronym: GENTLE:HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Virginia (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jill Howie Esquivel, PhD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21869
Record Dates: First submitted 2020-01-16; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: stretching; exercise; yoga; tele-health
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Educational Status; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Control Group (No Intervention): Education provided for optional use
- Gentle Stretching and Education (Experimental): Gentle Stretching for 60 minutes twice weekly for 6 months
  Interventions: Behavioral: Gentle Stretching and Education

INTERVENTIONS:
Behavioral: Gentle Stretching and Education — 60 minutes of gentle stretching twice weekly for 6 months
  Other Names: Exercise
  Arms: Gentle Stretching and Education

SUMMARY:
Despite scientific advances in treatment, patients with heart failure experience daily distressing symptoms and mortality rates are high. Although standard exercise improves numerous physical and psychological symptoms in heart failure patients, exercise participation rates are very low because of exercise barriers. Our research is aimed at understanding whether home-based gentle types of exercise such as yoga, delivered via video-conference, are beneficial in patients with heart failure. Challenging conventional strategies and breaking down barriers to care by testing new types of exercise delivered via tele-health (ipads) are urgently needed to improve the distressing symptoms that heart failure patients face daily.

DETAILED DESCRIPTION:
The over-arching goal of this research is to fill the substantial gap in knowledge about whether gentle forms of exercise will provide health benefits in patients with heart failure (HF). This gap is a particularly urgent problem as the prevalence and mortality rates for HF are rising. While medical therapy and standard exercise programs are known to decrease HF mortality and improve psychological outcomes, participation rates in standard exercise are low. Heart failure is a severe, life-limiting medical problem that affects millions of Americans and is the most common hospital discharge diagnosis in patients 65 and older. Patients with HF experience severe, distressing symptoms such as dyspnea and depression, along with co-morbid conditions that make standard exercise challenging. Therefore, lighter types of exercise, such as gentle stretching, may be particularly appealing and lead to higher exercise participation rates. Gentle stretching has been shown to improve blood pressure, breathlessness, and mood in patients with chronic diseases such as hypertension, lung disease, and depression, but few studies include patients with HF. Gentle stretching is an adaptable exercise that can be modified for co-morbid conditions such as arthritis, or symptoms, such as breathlessness. Our preliminary data show that short-term stretching is safe and feasible.

The goal of this study, GEtting iN To Light Exercise in Heart Failure: GENTLE-HF, is to test whether patients with stable HF will adhere to a long-term yoga exercise intervention, delivered via videoconferencing, using i-pads at home, compared to a health education group.

We will also test whether the intervention group has improvements in physical (endurance, balance, flexibility, strength) and psychological (depression, quality of life and self-care) function and HF severity biomarkers.

A sample of 100 adult HF patients will be recruited from the University of Virginia, Heart and Vascular Center Clinics and the University of California-John Muir. Yoga exercise participants will participate in 3 months of live, home-based, video-conference delivered, twice-weekly home yoga exercise classes, then 3 months of combined recorded and live exercise (6 months total) that enable transition to home exercise. The health education group participants will participate in 3 months of health education classes via ipad and then 3 months of reminders to complete symptom diaries. If effective, yoga exercise could be integrated into national guidelines for cardiac rehabilitation as a standard to improve distressing symptoms in patients with HF.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with reduced ejection fraction or Heart failure with preserved ejection fraction as seen by problem list in the EMR, is a patient in the heart failure clinic, or general cardiology clinic.
* ability to read, write and understand English;
* agree to participate and give informed consent;
* 19 years of age and older;
* telephone access;
* and NYHA class I-III with no changes in medications in 30 days (i.e. medical therapy is optimized).

Exclusion Criteria:

* are pregnant and/or breast feeding (self-reported)
* have a history of non-adherence with medications (as described by their provider or medical record);
* have had a hospitalization within the last 3 months for HF;
* have unstable angina; CABG, MI or biventricular pacemaker less than 6 weeks prior;
* have orthopedic impediments to stretching exercise; have severe COPD with a forced expiratory volume in one second less than 1 liter as measured by spirometry;
* have severe stenotic valvular disease;
* have a history of resuscitated sudden cardiac death without subsequent placement of an implantable cardioverter defibrillator;
* exercise more than 3 times weekly; currently engage in yoga at least 1 time per week;
* have cognitive impairment (as measured by the Mini-Cog)
* are living in a nursing home
* history of pulmonary arterial hypertension (PASP>60mmHg)
* other serious life-limiting co-morbidity, e.g. end stage cancer
* post-heart transplant (s/p OHT) or Left Ventricular Assist Device (LVAD)
* New York Heart Association Functional Class IV

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | 6 months
  Adherence will be determine by a class attendance rate of 80% to the intervention and the number of minutes of participation. A participation rate of 80% will be considered adherent.

SECONDARY OUTCOMES:
Cardiac Biomarkers | 6 months
  We will determine whether serum cardiac biomarkers of NT Pro-BNP and soluble ST-2 improve from baseline to after the intervention is complete.
Endurance | 6 months
  We will determine whether endurance improves using the 2 minute step test from baseline to after the intervention is complete.
Flexibility | 6 months
  We will determine whether hip flexibility improves using the sit and reach test from baseline to after the intervention is complete.
Upper body strength | 6 months
  We will determine whether upper body strength improves by measuring the number of arm curls completed in 30 seconds.
Lower body strength | 6 months
  We will measure quadricep strength by the number of times siting and standing in 30 seconds -participants are instructed to sit and then to stand as many times as possible in 30 seconds.
Balance | 6 months
  We will determine whether balance improves by measuring how many seconds a person can stand on 1 leg.
Heart Failure Somatic Perception Scale Questionnaire | 6 months
  This questionnaire measures symptoms of heart failure - The 18-item Somatic Perception Scale asks participants how much they are bothered by 18 symptoms of heart failure in the past week using 5 response options ranging from 0 (I did not have the symptom) to 5 (extremely bothersome). Scores are summed, with higher values indicating higher symptom burden. Scores range from 0-90 with higher values indicating higher symptom burden.
PROMIS questionnaire for depression | 6 months
  This questionnaire screens for symptoms of depression. The 8-item questionnaire assesses self-reported negative mood (sadness, guilt), views of self (self- criticism, worthlessness), and social cognition (loneliness, interpersonal alienation) in the past week. The questionnaire uses 5 response options ranging from 0 (never) to 5 (always). Scores are summed, with higher values indicating higher risk for depression. The total raw score is converted into a T-score. The T-score rescales the raw score into a standardized score. The final score is a standardized score with a mean of 50 and a standard deviation of 10.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 6 months
  This questionnaire measures quality of life in people with heart failure. This questionnaire is a 23-item, self- administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. In the KCCQ, a summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Overall scores are transformed to a range of 0-100, in which higher scores reflect better health status. There are summary scores within the KCCQ and the overall summary score is created by the mean of Physical Limitation Score, Total Symptom Score, Quality of Life Score, and Social Limitation Score.
The Resilience Scale | 6 months
  The Resilience Scale is a 25-item administered questionnaire that measures an individual's ability to adapt over time to stressors in life. Scores on the summated scale range from 25 to 175, with higher scores indicating higher resilience. All of the items are positively worded. Items are measured on a 7-point scale from 1(strongly disagree) to 7 (strongly agree). Responses are summed to produce a total score where a higher score indicates higher resilience.
Self-Care for Heart Failure Index Questionnaire (SCHFI) | 6 months
  The Self-Care for Heart Failure Index Questionnaire (SCHFI) is a 39-item measure of heart failure self-care. The items range from never (1) to always (5). There are 3 subscales: maintenance scale, symptom perception, confidence scale, and management scale. All of the scales are scored in the same way and a total score is not computed. Separate scores for each scale are computed separately.
  In general, to standardize a scale score, 1) determine the maximum possible scale score, 2) subtract the number of items from the possible score, and 3) divide 100 by that result to identify a constant for that scale. To score the scale, sum item responses, subtract the number of items answered, and multiply by the constant.The higher the score, the greater the ability to care for heart failure symptoms within each subscale.
The PROMIS Questionnaire for Anxiety | 6 months
  This questionnaire screens for symptoms of anxiety. The 8-item questionnaire assesses self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness) in the past week. The questionnaire uses 5 response options ranging from 1 (never) to 5 (always). To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40, with higher values indicating higher risk for anxiety. The total raw score is converted into a T-score. The T-score rescales the raw score into a standardized score. The final score is a standardized score with a mean of 50 and a standard deviation of 10. A score of 50 is the average for the United States general population.
The Pittsburgh Sleep Quality Index Questionnaire | 6 months
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in the older adult. It differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. The client self rates each of these seven areas of sleep. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale.
  A global sum of "5"or greater indicates a "poor" sleeper.
The FACIT-Sp Questionnaire for Spirituality | 6 months
  The 12-item Functional Assessment of Chronic Illness Therapy/Spiritual Well- being Scale (FACIT-Sp) is a measure of the religious/spiritual (R/S) components of quality of life (QoL). The questionnaire assessed the areas of spiritual well-being: meaning, peace and faith.
  Response for each item is assessed according to Likert scale 0-4 (0 - not in any event, 1 - small, 2 - somewhat, 3 - a lot, 4 - severe). The total score for each area is in the range 0-16, and total score of the whole scale is between 0 and 48. In all areas of the questionnaire higher scores indicated better quality of life, that is a spiritual well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Jill H Esquivel, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with investigators who request the dataset. No individual personal or HIPPA identifiers will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: When data are analyzed and for 5 years.

REFERENCES:
- [Background] Piepoli MF, Davos C, Francis DP, Coats AJ; ExTraMATCH Collaborative. Exercise training meta-analysis of trials in patients with chronic heart failure (ExTraMATCH). BMJ. 2004 Jan 24;328(7433):189. doi: 10.1136/bmj.37938.645220.EE. Epub 2004 Jan 16. PMID 14729656
- [Background] Pina IL, Apstein CS, Balady GJ, Belardinelli R, Chaitman BR, Duscha BD, Fletcher BJ, Fleg JL, Myers JN, Sullivan MJ; American Heart Association Committee on exercise, rehabilitation, and prevention. Exercise and heart failure: A statement from the American Heart Association Committee on exercise, rehabilitation, and prevention. Circulation. 2003 Mar 4;107(8):1210-25. doi: 10.1161/01.cir.0000055013.92097.40. No abstract available. PMID 12615804
- [Background] Flynn KE, Pina IL, Whellan DJ, Lin L, Blumenthal JA, Ellis SJ, Fine LJ, Howlett JG, Keteyian SJ, Kitzman DW, Kraus WE, Miller NH, Schulman KA, Spertus JA, O'Connor CM, Weinfurt KP; HF-ACTION Investigators. Effects of exercise training on health status in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1451-9. doi: 10.1001/jama.2009.457. PMID 19351942
- [Background] Blumenthal JA, Babyak MA, O'Connor C, Keteyian S, Landzberg J, Howlett J, Kraus W, Gottlieb S, Blackburn G, Swank A, Whellan DJ. Effects of exercise training on depressive symptoms in patients with chronic heart failure: the HF-ACTION randomized trial. JAMA. 2012 Aug 1;308(5):465-74. doi: 10.1001/jama.2012.8720. PMID 22851113
- [Background] Kulcu DG, Kurtais Y, Tur BS, Gulec S, Seckin B. The effect of cardiac rehabilitation on quality of life, anxiety and depression in patients with congestive heart failure. A randomized controlled trial, short-term results. Eura Medicophys. 2007 Dec;43(4):489-97. PMID 18084172
- [Background] WRITING COMMITTEE MEMBERS; Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):e240-327. doi: 10.1161/CIR.0b013e31829e8776. Epub 2013 Jun 5. No abstract available. PMID 23741058
- [Background] Yates BC, Pozehl B, Kupzyk K, Epstein CM, Deka P. Are Heart Failure and Coronary Artery Bypass Surgery Patients Meeting Physical Activity Guidelines? Rehabil Nurs. 2017 May-Jun;42(3):119-124. doi: 10.1002/rnj.257. PMID 29203953
- [Background] Park LG, Schopfer DW, Zhang N, Shen H, Whooley MA. Participation in Cardiac Rehabilitation Among Patients With Heart Failure. J Card Fail. 2017 May;23(5):427-431. doi: 10.1016/j.cardfail.2017.02.003. Epub 2017 Feb 14. PMID 28232047
- [Background] Rengo JL, Savage PD, Barrett T, Ades PA. Cardiac Rehabilitation Participation Rates and Outcomes for Patients With Heart Failure. J Cardiopulm Rehabil Prev. 2018 Jan;38(1):38-42. doi: 10.1097/HCR.0000000000000252. PMID 28671938
- [Background] Blackburn GG, Foody JM, Sprecher DL, Park E, Apperson-Hansen C, Pashkow FJ. Cardiac rehabilitation participation patterns in a large, tertiary care center: evidence for selection bias. J Cardiopulm Rehabil. 2000 May-Jun;20(3):189-95. doi: 10.1097/00008483-200005000-00007. PMID 10860201